CLINICAL TRIAL: NCT02351518
Title: Cerebral Autoregulation and Vasospasm in Patients With Traumatic Brain Injury
Brief Title: Cerebral Autoregulation and Vasospasm in Patients With TBI
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Deborah Stein, Professor, Department of Surgery, University of Maryland , Chief of Trauma R Adams Cowley Shock Trauma Center, University of Maryland, Baltimore
Other Study IDs: HP-00062723
Record Dates: First submitted 2015-01-19; First posted 2015-01-30 (Estimated); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Tbi; Vasospasm; Cerebral Ischemia; Cerebral Infarct
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Ischemia; Cerebral Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention — There will be no interventions in this study

SUMMARY:
Traumatic brain injury (TBI) affects 1.5 million patients per year in the United States, resulting in more than 50,000 deaths and more than 230,000 hospitalizations annually. Approximately 90,000 of these patients will suffer permanent impairment and more than half will experience short-term disability.

Secondary injury processes play a critical role in the development of ischemia after trauma to the central nervous system and occur hours-to-days after the primary insult. Ischemia can lead to cerebral infarction or stroke. Ischemia has been described as the single most important secondary insult and has been identified histologically in approximately 90% of patients who die following closed head injury. Several factors resulting in post-traumatic cerebral ischemia have been identified: increased intracranial pressure (ICP), systemic arterial hypotension, and cerebral vasospasm. Cerebral vasospasm has been described as a sustained arterial narrowing. Clinically, the onset of new or worsening neurological symptoms is the most reliable indicator of cerebral vasospasm following a ruptured cerebral aneurysm. However, cerebral vasospasm is often unrecognized in patients suffering from moderate to severe TBI. These patients frequently have altered mental status due to the primary brain injury. In addition, they require narcotics for their pain and paralytics and/or sedatives while on a mechanical ventilator for airway protection. Thus, relying on the neurological exam to observe deteriorating neurological signs consistent with post-traumatic vasospasm (PTV) is reliable. While the etiology and outcome of patients with vasospasm secondary to ruptured aneurysm is well documented, the clinical significance of PTV after TBI is unknown. A better understanding of the role of cerebral autoregulation in the development of cerebral vasospasm could provide the answer. This proposal is for a pilot observational study describing the association of the impairment of cerebral autoregulation as measured by near infrared spectroscopy (NIRS) with the development of clinically significant vasospasm in patients with moderate to severe TBI. The information will serve as preliminary data for further study.

DETAILED DESCRIPTION:
Primary Objectives: 1. To determine if impaired cerebral autoregulation as measured by NIRS is associated with clinically significant vasospasm in patients with moderate to severe TBI; 2. To determine the sensitivity and specificity of NIRS in detecting clinically significant vasospasm with Transcranial Doppler (TCD) ultrasound followed by CT brain angiography and diffusion-weighted brain MRI as the gold standard . Secondary Objectives: 1. To determine the relationship between impaired cerebral autoregulation and outcomes; 2. To determine the relationship between impaired cerebral autoregulation, clinically significant vasospasm and outcomes

Clinical observations The subject will be continuously monitored with INVOS NIRS system within the first 24 hours after admission up to 7 days while the subject is still in the STC. If decreased cerebral oxygenation is detected by NIRS, TCDs will be offered to the family and considered part of routine clinical care. If vasospasm is detected by TCD, CT brain angiography will be offered to the family for angiographic confirmation and considered part of routine clinical care. If vasospasm is confirmed by CT brain angiography, diffusion-weighted MRI will be offered to the family to evaluate for cerebral ischemia/infarction and considered part of routine clinical care.

Laboratory evaluations All patients will have at least twice daily measurements of serum electrolytes, blood counts, arterial blood gases, and coagulation profile as per our standard of care. Culture results will be recorded. No tests or procedure will be ordered for research purposes only.

Patient Management All enrolled patients will be admitted to the Neurotrauma Critical Care Unit (NTCC) and be jointly managed by the Trauma, Critical Care and Neurosurgical services. All patients will be managed utilizing the STC Institutional Severe Traumatic Brain Injury Management Algorithm which is based on the Brain Trauma Foundation Guidelines for the Management of Severe Traumatic Brain Injury. Other consults will be obtained as clinically indicated.

Questionnaires / Assessment tools Functional outcome using the Extended Glasgow Outcome Scale (GOS-E) will be assessed in the STC Outpatient Clinic as part of their standard of care. An early functional outcome assessment will be obtained if the GOS-E form is completed at the STC Outpatient Clinic within 6 weeks post hospital discharge day. A mid functional outcome assessment will be obtained if the GOS-E form is completed at the STC Outpatient Clinic 6 weeks to 3 months post hospital discharge day. A late functional outcome assessment will be obtained if the GOS-E form is completed at the STC Outpatient Clinic 3 months to 6 months post hospital discharge day. Finally, a very late functional outcome assessment will be obtained if the GOS-E form is completed at the STC Outpatient Clinic more than 6 months post-hospital discharge day.

STATISTICAL CONSIDERATIONS / ANALYSIS OF DATA The goal of this pilot study is to determine if impaired cerebral autoregulation as measured by NIRS is associated with the development of clinically significant vasospasm in patients with moderate to severe TBI. By enrolling 100 patients in the study, it is expected to estimate the correlation to within 0.098 with a probability of at least 95%. In this study, all primary and secondary outcomes may be classified into two categories: binary and continuous. In the first step, quantitative descriptive statistics will be used initially to study the characteristics of patients and the association between clinical outcomes (e.g. vasospasm) and various demographic and clinicopathologic variables such as age, gender and injury severity scores. For binary data, chi-square and Fisher's exact tests will be used to identify differences. For continuous variables, t-tests and analysis of variance (ANOVA) will be used to determine the significant association. These univariate tests will be done at a significance level of 0.05. In addition to constructing 95% confidence interval for the correlation of impaired cerebral autoregulation as measured by NIRS and clinically significant vasospasm, the investigators will also explore potential risk factors associated with impaired cerebral autoregulation and impaired cerebral autoregulation associated with vasospasm. To this end, the correlation will be analyzed using the logistic regression model with various demographic and clinicopathologic variables as independent variables. The stepwise regression procedure will be used for identifying potential risk factors for the incidence of vasospasm. To evaluate the validity of NIRs as an assessment method of vasospasm, the investigators will measure the agreement between TCD and NIRS by using kappa statistics.

ELIGIBILITY:
Inclusion Criteria:

* 15 years of age and greater
* Motor Glasgow Coma Score (GCS) < 6 within approximately 24 hours of admission
* Head AIS > 2

Exclusion Criteria:

* Motor GCS >5
* Determination of non-survivability on admission
* Non-English speakers
* Prisoners that are on parole or probation
* Active duty military
* Pregnant patients

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients aged 15 years and older, presenting with a motor score of <6 and thought to have TBI due to a mechanism of injury, will undergo screening with head computed tomography (CT). Admission CT will be interpreted by an attending radiologist to determine Head Abbreviated Injury Score (AIS) score. If the AIS score by CT is > 2, the patient will be eligible for the study. Patients determined by neurosurgery to have a non-survivable TBI on admission will be excluded given the poor likelihood of completion of the study protocol.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-11; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Functional Outcome as assessed by the Glasgow Functional Outcome-Extended | within 12 months post hospital discharge

SECONDARY OUTCOMES:
Mortality | within 30 days
Hospital Length of Stay | within 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Stein, MD, MPH, Principal Investigator — Professor of Surgery, Department of Surgery, Chief of Trauma R Adams Cowley Shock Trauma Center
Locations (1):
- R Adams Cowley Shock Trauma Center, University of Maryland Medical Center, Baltimore, Maryland, United States